CLINICAL TRIAL: NCT00053560
Title: A Randomized, Double-Blind, Multi-Center, Placebo- Controlled Study to Assess Prevention of Bone Loss by Treatment With GL701 (Prestara) in Women With Systemic Lupus Erythematosus Receiving Treatment With Glucocorticoids
Brief Title: To Assess Prevention of Bone Loss in Women With Lupus Receiving Treatment With Glucocorticoids
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genelabs Technologies (Industry)
Responsible Party: Kenneth E. Schwartz, MD/Vice President, Medical Affairs, Genelabs Technologies, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GL02-01
Record Dates: First submitted 2003-01-30; First posted 2003-02-03 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2004-11

CONDITIONS: Lupus
Keywords: lupus; systemic lupus erythematosus; SLE; bone loss; DHEA
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Bone Diseases, Metabolic | interventions — Dehydroepiandrosterone; GL-701

INTERVENTIONS:
Drug: Prasterone (GL701)

SUMMARY:
The purpose of this clinical trial is to study the effects of GL701 on bone mineral density in women with active systemic lupus erythematosus (SLE) who are also receiving treatment with glucocorticoids (e.g., prednisone).

ELIGIBILITY:
INCLUSION CRITERIA

* Women at least 18 years of age.
* Meet ACR criteria for diagnosis of SLE.
* Concomitant treatment with prednisone at a dose of ≥5 mg/day over the last 30 days prior to Screening visit.
* Cumulative history of oral glucocorticoid use for at least 6 months over the last year prior to the Screening Visit (the 6 months do not have to be consecutive).
* Patient has lumbar spine and proximal femur anatomy suitable for measurement by DXA with at least 3 evaluable vertebrae from L1 to L4.
* SLEDAI ≥3 at the Qualifying Visit.
* Women of child-bearing potential must have a negative serum pregnancy test (at the Screening Visit) and agree to use a reliable form of birth control while participating in the study.
* Patient is fully ambulatory.
* Patient has read and signed an Informed Consent Form.

EXCLUSION CRITERIA

* History of breast cancer or malignancy of the reproductive tract organs.
* History of any other cancers unless no evidence of disease for 5 years.
* History of endometrial hyperplasia.
* End stage renal disease or receiving hemodialysis treatment.
* Any disease or condition that would preclude the accurate measurement of bone mineral density of the lumbar spine or proximal femur by dual X-ray absorptiometry.
* A T-score of less than or equal to - 2.5 of the L-spine or proximal femur at Screening DXA assessment.
* Unstable cardiac disease.
* Conditions causing bone loss such as hyperparathyroidism, Cushing's disease, thyrotoxicosis, chronic diarrheal state or malabsorption, renal tubular acidosis, or anorexia nervosa.
* Significant hepatic disease (i.e., cirrhosis).
* Body mass index > 35 kg/m2 or weight >300 lbs.
* Patients who are pregnant or breast feeding.
* Patients who require glucocorticoids by an alternate day dosing schedule.
* Known hypersensitivity to DHEA, or the inactive ingredients used in the GL701 formulation (cornstarch, lactose, magnesium stearate).
* Known medical contraindication or hypersensitivity to Calcium/Vitamin D.
* Participation in any prior DHEA or GL701 study.
* Use of investigational agents within 30 days of the Screening Visit or 10 half-lives of the agent.
* Any condition which in the Investigator's or Sponsor's opinion is sufficient to prevent adequate compliance with the study or likely to confuse follow-up evaluation (e.g., alcoholism, drug addiction, acute withdrawal from chemical dependency, psychiatric disease).
* The patient is taking or has taken one of the medications listed below:

ANTIRESORPTIVES:

* Use of calcitonin within 30 days prior to Screening Visit.
* Fluorides > 1 mg/day at any time prior to the study.
* Strontium at pharmacologic dose at any time.

BISPHOSPHONATE USE as follows:

* Any use within 90 days prior to the Screening Visit.
* ≥ 2 weeks of use in the last year prior to the Screening Visit.
* ≥ 3 months of use in the last 2 years prior to the Screening Visit.
* ≥ 1 intravenous dose over the last 2 years prior to the Screening Visit.
* ≥ 6 months of life-time exposure prior to the Screening Visit.

ESTROGENIC STEROIDS (Except for oral contraceptives):

* Estrogenic steroids (HRT) within 60 days of the Screening Visit.
* Selective estrogen receptor modulator (raloxifene) within 60 days of the Screening Visit.

OTHER HORMONES:

* Parathyroid hormone (PTH) within six months of the Screening Visit.
* Use of any androgens, including prescription or nutritional supplement DHEA, within 30 days of the Screening Visit.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155
Dates: Start 2002-12; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Locations (26):
- United States (25):
  - University of Arizona, Tucson, Arizona
  - Wallace Rheumatic Study Center, Los Angeles, California
  - Peng T Fan, MD & Wonil Lee, MD Partnership, North Hollywood, California
  - Lifestyles Health Science Center, Rancho Mirage, California
  - University of California San Diego, San Diego, California
  - East Bay Rheumatology Group, San Leandro, California
  - Center for Rheumatology, Immunology and Arthritis, Fort Lauderdale, Florida
  - Rheumatology Associates of Central Florida, Orlando, Florida
  - Tampa Medical Group, P.A., Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - St. John's Medical Research Group, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - SUNY Downstate Medical Center, Brooklyn, New York
  - North Shore University Hospital, Division of Rheumatology, Manhasset, New York
  - Albert Einstein Medical School, The Bronx, New York
  - Oklahoma Center for Arthritis Therapy, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas, Medical Branch, Galveston, Texas
  - Sentara Medical Group DBA, Virginia Beach, Virginia
  - Seattle Rheumatology Associates, Seattle, Washington
- Immunology/Rheumatology Instituto Nacional de Ciencias Medicas y Nutricion, S.Z., Mexico City, Mexico

REFERENCES:
- [Derived] Sanchez-Guerrero J, Fragoso-Loyo HE, Neuwelt CM, Wallace DJ, Ginzler EM, Sherrer YR, McIlwain HH, Freeman PG, Aranow C, Petri MA, Deodhar AA, Blanton E, Manzi S, Kavanaugh A, Lisse JR, Ramsey-Goldman R, McKay JD, Kivitz AJ, Mease PJ, Winkler AE, Kahl LE, Lee AH, Furie RA, Strand CV, Lou L, Ahmed M, Quarles B, Schwartz KE. Effects of prasterone on bone mineral density in women with active systemic lupus erythematosus receiving chronic glucocorticoid therapy. J Rheumatol. 2008 Aug;35(8):1567-75. Epub 2008 Jul 15. PMID 18634158